CLINICAL TRIAL: NCT03897530
Title: Flavored Tobacco Product Regulation: Behavioral Economic Demand, Visual Attention, and Flavored Tobacco Product Availability
Brief Title: Experimental Tobacco Marketplace in Regulating Flavored Tobacco Products in Menthol Cigarette Smokers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: I 75418; R03CA228930 (NIH)
Record Dates: First submitted 2019-03-26; First posted 2019-04-01 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (Experimental): During the session, participants are presented with randomly ordered conditions: menthol cigarettes and five flavored e-cigarettes (menthol/mint, fruits, sweets, alcohol, snacks/meals), menthol cigarettes and both unflavored and tobacco-flavored e-cigarettes, non-menthol cigarettes and five flavored e-cigarettes, and non-menthol cigarettes and both unflavored and tobacco-flavored e-cigarettes. Participants' visual attention is evaluated by eye-tracking equipment.
  Interventions: Behavioral: Smoking Cessation Intervention; Other: Functional Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Smoking Cessation Intervention — View and purchase hypothetical tobacco products during four distinctly different ETM
Other: Functional Assessment — Visual attention is evaluated via eye-tracking equipment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial uses an Experimental Tobacco Marketplace to study the purchase of tobacco products in menthol cigarette smokers. Determining the level of substitutability of both flavored and unflavored/tobacco flavored e-cigarettes when menthol cigarettes are available and unavailable can help determine if a flavor ban (of either menthol cigarettes and/or flavored e-cigarettes) will lead to smoking cessation and/or harm reduction. A greater understanding of tobacco product purchasing could help inform possible regulatory actions by the Food and Drug Administration.

DETAILED DESCRIPTION:
Participants view and purchase hypothetical tobacco products during four distinctly different Experimental Tobacco Marketplace (ETM) conditions. During the session, participants are presented with these randomly ordered conditions: menthol cigarettes and five flavored e-cigarettes (menthol/mint, fruits, sweets, alcohol, snacks/meals), menthol cigarettes and both unflavored and tobacco-flavored e-cigarettes, non-menthol cigarettes and five flavored e-cigarettes, and non-menthol cigarettes and both unflavored and tobacco-flavored e-cigarettes. Participants' visual attention is evaluated by eye-tracking equipment.

ELIGIBILITY:
Inclusion Criteria:

* Menthol cigarette smokers who report smoking a brand that has a non-menthol equivalent.
* Residing in Western New York.
* Voluntarily provide informed consent to participate in the study.

Exclusion Criteria:

* Any known history of macular degeneration, glaucoma, cataracts, eye implant, permanently dilated pupils or the use of a screen reader/magnifier.
* The following special populations will not be included:

  * Adults unable to consent
  * Individuals who are not yet adults (infants, children, teenagers)
  * Prisoners
  * Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Cessation of Menthol flavored cigarettes | At the time of the session , assessed up to 15 months
  Number of flavored cigarettes purchased inThe Experimental Market Place (ETM) will be used to track tobacco purchase behaviors
Eye tracking metrics | At the time of the session , assessed up to 15 months
  the interaction of type of cigarette available (menthol versus non-menthol) and type of e-cigarette available (flavors versus unflavored and tobacco), will employ a 2 X 2 repeated measures ANOVA with post-hoc Bonferroni tests to evaluate the outcomes of Q0 (derived initial consumption without cost constraints), α (demand elasticity), the substitution levels, and the eye-tracking metrics.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Quisenberry, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT03897530/ICF_000.pdf